CLINICAL TRIAL: NCT01922648
Title: Analysis of the Immune Response to Respiratory Syncytial Virus (RSV) Exposure in a Paediatric Population
Brief Title: RSV Observational Study 2
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/01
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV; Immune response; Paediatric
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 2-4 months: Infants aged between 2 and 4 months (Group 1), who have not yet been exposed to RSV
  Interventions: Procedure: Blood sample
- 6 - 12 months: Infants aged between 6 and 12 months (Group 2), who will have had exposure to one single RSV season in the winter of 2011/12
  Interventions: Procedure: Blood sample
- 3 - 6 years: Children aged between 3 and 6 years (Group 3), who have been exposed to RSV over several winter seasons
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — An extra volume of blood is obtained, with prior consent, when phlebotomy is required for another unrelated clinical reason.

SUMMARY:
Respiratory Syncytial Virus (RSV) is a virus that causes chest infections. It is the single most important cause of severe respiratory illness in infants and young children, and severe RSV infection early in life is associated with an increased risk of later developing asthma. RSV also causes severe disease in elderly and immune-compromised adults, and the amount of RSV disease in the elderly is similar to that from seasonal flu. The virus is transmitted in the secretions of the upper respiratory tract of infected individuals and by contact with contaminated surfaces (such as toys). Hospital outbreaks, especially on paediatric and neonatal wards, are not uncommon.

Infection by RSV does not develop a natural long-lasting protection against re-infection (like, for example, measles does). In the USA nearly all children by 24 months of age have been infected at least once with RSV, and about half will have experienced two infections. There is no effective anti-viral drug to treat an infection and the only way of managing cases of severe infection is through supporting organs, such as the lungs, to withstand and recover from the illness.

There remains a real need to develop an effective vaccine to prevent severe infections caused by RSV. A better understanding of the way the immune system responds to RSV in children would aid the development of such a vaccine.

The purpose of this study is to increase our understanding of how the immune system responds to RSV. Only limited data is available on some important components of the immune response and this study is designed to measure these in more detail. This is done using a single blood sample.

A total of 35 children are anticipated to be recruited to this study, at ages when we expect to see differences in the immune response to RSV;

* 5 infants aged between 2 and 4 months (Group 1), who have not yet been exposed to RSV
* 20 infants aged between 6 and 12 months (Group 2), who will have had exposure to one single RSV season in the winter of 2011/12
* 10 children aged between 3 and 6 years (Group 3), who have been exposed to RSV over several winter seasons

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian is willing and able to give informed consent for participation in the study
* Age suitable for Group 1, 2 or 3 as defined in above (Section 6.2)
* Delivery at 36 weeks gestation or later
* Having a blood sample for clinical reasons

Exclusion Criteria:

* Parent or guardian unable or unwilling to give informed consent for participation in the study
* Any impaired function of the immune system, by medication or pathological process, which could augment or impair the immune response to RSV
* Concurrent acute or chronic infection
* Any chronic illness which, in the opinion of the Investigator, may lead to incorrect or inaccurate immunology data
* History of immunoprophylaxis with Palivizumab
* Delivery prior to 36 weeks gestation

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants aged 2-4 months inclusive Infants aged 6-12 months inclusive Children aged 3-6 years inclusive
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-06; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To assess the induction of RSV-specific immune responses in blood following natural exposure | one year
  The following assays characterise the primary objective:
  * Anti-RSV antibody concentration and neutralisation capacity
  * T-cell immune responses

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hopsitals NHS Trust, Oxford, United Kingdom